CLINICAL TRIAL: NCT01348529
Title: Internet-based Cognitive Behavior Therapy for Obsessive Compulsive Disorder: A Pilot Study
Brief Title: Internet Cognitive Behavior Therapy (CBT) for Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Christian Rück, MD, PhD, Study Principal Investigator, Karolinska Institutet, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCDP1
Record Dates: First submitted 2010-11-08; First posted 2011-05-05 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2010-09

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; CBT; Reducing OCD symptoms
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet CBT (Experimental): Internet-delivered cognitive behavioral therapy with therapist support.
  Interventions: Behavioral: Internet CBT

INTERVENTIONS:
Behavioral: Internet CBT — Internet-delivered cognitive behavioral therapy with therapist support.

SUMMARY:
The main aim of this study is to test whether cognitive behavior therapy could be effective in treating obsessive compulsive disorder. Here, the investigators test the in group effects of a 15 week long treatment delivered via the Internet for residents in Stockholm County.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Obsessive compulsive disorder according to the DSM criteria
* Be at least 18 years old
* YBOCS >7

Exclusion Criteria:

* other primary diagnosis
* substance abuse,
* psychosis,
* bipolar disorder,
* suicidal ideation,
* adjusted pharmacological treatment the last two months
* current psychological treatment for OCD,
* been treated with CBT the last two years,
* serious somatic disease,
* Y---BOCS>31
* hoarding as primary OCD subtype

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of obsessions and compulsions after 15 weeks and 6 months after treatment. | Psychiatrist visit at baseline, after 15 weeks of treatment and 6 months after treatment.
  Yale Brown Obsessive Compulsive Scale (Y-BOCS)

SECONDARY OUTCOMES:
Change from Baseline of cost data after 15 weeks and 6 months after treatment. | Self-ratings at baseline, after 15 weeks of treatment and 6 months after treatment.
  "Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry". In this questionnaire, patients register their monthly health care consumption (e.g. GP visits) as well as time spent in informal health enhancing activities (e.g. self-help groups and informal care from friends). In addition, work loss and work cutback both at work and in the domestic realm is measured.
Change from Baseline of depressive symptoms after 15 weeks and 6 months after treatment. | Sel-ratings at baseline, after 15 weeks of treatment and 6 months after treatment.
  The Montgomery Åsberg Depression Rating Scale
Change from Baseline of obsessions and compulsions after 15 weeks and 6 months after treatment. | Self-ratings at baseline, after 15 weeks of treatment and at 6 months after treatment.
  Obsessions and Compulsions Inventory Revised
Change from Baseline of quality of life after 15 weeks and 6 months after treatment | Self-ratings at baseline, after 15 weeks of treatment and at 6 months after treatment.
  EuroQol
Change from Baseline of quality of life after 15 weeks and 6 months after treatment | Self-ratings at baseline, after 15 weeks of treatment and at 6 months after treatment.
  Quality of life inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Internetpsykatrienheten, M46, Psykiatri sydväst, Stockholm, Sweden

REFERENCES:
- [Result] Andersson E, Ljotsson B, Hedman E, Kaldo V, Paxling B, Andersson G, Lindefors N, Ruck C. Internet-based cognitive behavior therapy for obsessive compulsive disorder: a pilot study. BMC Psychiatry. 2011 Aug 3;11:125. doi: 10.1186/1471-244X-11-125. PMID 21812991
- See also: Related Info — http://www.internetpsykiatri.se